CLINICAL TRIAL: NCT03593161
Title: The Effect of Humor Therapy on Perceived Distress After Allogeneic Stem Cell Transplantation
Brief Title: Humor Therapy and Distress After Allogeneic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Deutsche José Carreras Leukämie-Stiftung (Unknown); Staburo GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DJCLS 26R/2017
Record Dates: First submitted 2018-06-11; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: stem cell transplantation; allogeneic; humor therapy; distress; supportive care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Humor therapy (Experimental): After baseline assessment (before start of conditioning), patients assigned to the experimental study arm will receive the standard psychosocial care plus weekly clown visits over the course of their inpatient stay for allogeneic stem cell transplantation.
  Interventions: Behavioral: Humor therapy
- Treatment as usual (No Intervention): Patients assigned to the control arm will receive the standard psychosocial care over the course of their inpatient stay for allogeneic stem cell transplantation.

INTERVENTIONS:
Behavioral: Humor therapy — Clown visits
  Arms: Humor therapy

SUMMARY:
This research study evaluates the impact of a humor intervention on distress (primary outcome), hope, depressive symptoms, anxiety, and pain (secondary outcomes) in patients undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT).

DETAILED DESCRIPTION:
Patients undergoing allo-HSCT often experience substantial psychological distress during hospitalization and after discharge. Research in pediatric patients with cancer as well as geriatric patients suggests that psychosocial burden might be decreased by humor therapy. Studies addressing the impact of humor therapy in adult patients with cancer are lacking.

This randomized controlled trial primarily aims at assessing the effect of therapeutic humor on global distress in patients during their hospital stay for allo-HSCT. In addition, the study investigates hope, depressive symptoms, anxiety, and pain as secondary outcomes. The outcomes are measured via questionnaires.

Study results may be beneficial for patients who experience distress during hospitalization for allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission for allogeneic transplantation at the University Medical Center Hamburg-Eppendorf

Exclusion Criteria:

* Insufficient German language skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Distress | Change from baseline (before start of conditioning) to 4 weeks after allogeneic stem cell transplantation (days +7, +14, +21 and +28)
  Measured with the Distress Thermometer (DT): Brief screening instrument to assess the level of perceived distress in patients with cancer (11-point scale ranging from 0 = no distress to 10 = extreme distress)

SECONDARY OUTCOMES:
Hope | Change from baseline (before start of conditioning) to 4 weeks after allogeneic stem cell transplantation (days +7, +14, +21 and +28)
  Measured with the Herth Hope Index (HHI): Short self-report instrument for the measurement of hope in clinical oncological care (12 items, 4-point Likert scale ranging from 1 = strongly disagree to 4 = strongly agree)
Depressive symptoms | Change from baseline (before start of conditioning) to 4 weeks after allogeneic stem cell transplantation (days +14 and +28)
  Measured with the Patient Health Questionnaire-9 (PHQ-9): Short self-report instrument to assess the severity of depressive symptoms (9 items, 4-point Likert scale ranging from 0 = not at all to 3 = nearly every day)
Anxiety symptoms | Change from baseline (before start of conditioning) to 4 weeks after allogeneic stem cell transplantation (days +14 and +28)
  Measured with the Generalized Anxiety Disorder Scale-7 (GAD-7): Short self-report instrument to assess the severity of anxiety symptoms (7 items, 4-point Likert scale ranging from 0 = not at all to 3 = nearly every day)
Pain intensity measured with the Numerical Rating Scale (NRS) | Change from baseline (before start of conditioning) to 4 weeks after allogeneic stem cell transplantation (days +7, +14, +21 and +28)
  Measured with the Numerical Rating Scale (NRS): Brief screening instrument to assess pain intensity (11-point scale ranging from 0 = no pain to 10 = worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus M. Kröger, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Department of Stem Cell Transplantation
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany